CLINICAL TRIAL: NCT02999932
Title: Effect of Low vs High Peripheral Oxygen Saturation (SpO2) Directed Oxygen Therapy on Mortality Among Critically Ill Patients
Brief Title: Peripheral Oxygen Saturation (SpO2) Directed Oxygen Therapy
Acronym: POSDOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Principal Investigator, Xiaobo Yang, MD, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WuhanUHICU201701
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low SpO2 group (Experimental): SpO2 90-95%, with FiO2 as low as possible.
  Interventions: Other: SpO2 directed oxygen therapy
- High SpO2 group (Active Comparator): SpO2 96-100%, with FiO2 no lower than 30%.
  Interventions: Other: SpO2 directed oxygen therapy

INTERVENTIONS:
Other: SpO2 directed oxygen therapy — Oxygen therapy was administered to achieve targeted SpO2.

SUMMARY:
Investigators hypothesized that a relative low SpO2 directed oxygen therapy would reduced the mortality in patients staying longer than 72 hours in ICUs.

DETAILED DESCRIPTION:
In fear of harmful effect of hypoxia, oxygen therapy is commonly used, especially in critically ill patients in intensive care units (ICUs). However, hyperoxia can be harmful too. Examples are myocardial infarction (MI) patients and patients resuscitated to return of spontaneous circulation after cardiac arrest. In Air Versus Oxygen in Myocardial Infarction (AVOID) trial, Meyhoff and colleagues proved hyperoxia caused more cardiac injury in patients with ST-elevation MI but without hypoxia. Kilgannon and colleagues found that arterial hyperoxia following resuscitation from cardiac arrest were associated with increased in-hospital mortality, and a pulse oxygen saturation (SpO2) of 94-98% was recommended.

Recently, Panwar and colleagues found that compared to liberal oxygen strategy (SpO2 ≥96%), conservative oxygen strategy (SpO2 of 88%-92%) was feasible in patients receiving invasive mechanical ventilation. Girardis and colleagues found control oxygen therapy (targeting SpO2 of 94%-98% or PaO2 of 70-100mmHg) resulted lower ICU mortality than conventional oxygen therapy (SpO2 ≥97%) in the randomized clinical trial called Oxygen-ICU. However, the Oxygen-ICU trial was single-centered, early-terminated with only 480 patients included and led to an unplanned interim analysis. In this larger multicenter trial, investigators hypothesized that a relative low SpO2 directed oxygen therapy was safe and would reduced the 28-day mortality in patients staying longer than 72 hours in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older and admitted into ICU, with expected stay in ICU more than 72 hours or longer.

Exclusion Criteria:

* under 18 years old, expected stay in ICU less than 72 hours, unconsented inclusion, ICU readmission, patients with acute exacerbation of chronic obstruction disease, patients with severe acute respiratory distress syndrome (defined as PaO2/FiO2 ≤ 100mmHg and PEEP ≥10cmH2O), decision to withhold life-sustaining treatment, physician forgetting to screen during 12 hours after admission, pregnancy, patients with acute myocardial infarction, paraquat poisoning and patients on extracorporeal membrane oxygenation (ECMO) or planned to be on ECMO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1706 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  Death within 28 days after inclusion

SECONDARY OUTCOMES:
ventilator-free time | 14 days
  Hours free from ventilator
RRT-free time | 14 days
  Hours free from renal replacment therapy

CONTACTS AND LOCATIONS:
Overall Officials: Shiying Yuan, MD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (13):
- China (13):
  - Department of critical care medicine，Luoyang Central Hospital Affiliated to ZhengZhou University, Luoyang, Henan
  - Department of critical care medicine，Xinyang Central Hospital, Xinyang, Henan
  - Department of critical care medicine, Henan Provincial People's Hospital, Zhengzhou, Henan
  - Department of critical care medicine, The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Department of critical care medicine，Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Department of critical care medicine, Renmin Hospital of Shiyan City, Shiyan, Hubei
  - Department of critical care medicine, Taihe Hospital, Shiyan, Hubei
  - Department of critical care medicine, The Central Hospital of Wuhan, Wuhan, Hubei
  - Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of critical care medicine，Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Intensive Care Unit, Hubei Cancer Hospital, Wuhan, Hubei
  - Department of critical care medicine, Xiangyang No.1 People's Hospital, Affiliated Hospital of Hubei University of Medicine, Xiangyang, Hubei
  - Department of critical care medicine, XiangYang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science, Xiangyang, Hubei

IPD SHARING:
Plan to Share IPD: Undecided